CLINICAL TRIAL: NCT04403607
Title: Cardiovascular and Pulmonary Imaging in SARS-CoV-2: A Study of the Heart, Lungs and Wellbeing After COVID-19.
Brief Title: Cardiac Imaging in SARS-CoV-2 (COVID-19)
Acronym: CISCO-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN20ID164
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be stored for biomarker analyses including DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Patients with confirmed COVID-19 meeting the eligibility criteria specified in the protocol.
- Control: COVID-19 negative. Age/sex matched to the COVID-19 cohort. Age range 40-80 years. At least one cardiovascular risk factor by ASSIGN criteria.

SUMMARY:
One-in-four patients with COVID-19 pneumonia develop life-threatening heart problems. Through cardiovascular imaging and biomarkers analyses this study aims to evaluate whether COVID-19 infection results in heart injury. The investigators will also investigate which patients are at risk of heart injury as a result of COVID-19 and why only some patients suffer heart problems as a consequence of the infection. The study will also assess multisystem involvement including the lungs and kidneys.

DETAILED DESCRIPTION:
Our study is supported through the Chief Scientist Office Rapid Research in Covid-19 (RARC-19) programme. Our study will clarify the pathogenesis of cardiopulmonary injury, notably endotypes of myocardial injury including myocarditis, in patients with COVID-19.

The study involves a prospective, observational, multicentre, longitudinal cohort design.The investigators aim to minimise selection bias by adopting consecutive screening of all-comers hospitalised with COVID-19 and the eligibility criteria are broad. For example, severe renal dysfunction is not an exclusion criterion. The sample size is 180 patients enrolled at baseline with 160 attending for the primary outcome evaluation (cardiac imaging) at 28 days post-discharge. The investigators will use advanced cardiovascular imaging to identify the number (proportion) of patients with myocardial inflammation (myocarditis) that is sub-clinical (i.e. not diagnosed) or clinically overt. Cardiovascular MRI and CT coronary angiography will provide a comprehensive examination one month after discharge is intended to detect persisting cardiovascular complications and diagnose clinical endotypes. The investigators aim to clarify the pathological significance of serial changes in circulating troponin, NTproBNP and renal function. By correlating the MRI findings with troponin I and other measures of cardiovascular injury, such as NTproBNP, our results will inform care pathways that use these blood tests to guide the management of patients with COVID-19. Correlation of imaging findings with baseline clinical information, biomarkers, patient reported outcome measures and well-being in the longer term will help to clarify the clinical significance of cardiovascular complications in COVID-19. Since the design is observational, an interim analysis may be undertaken with the timing informed by the enrolment rate.

Longer term follow-up will include a 5-year visit, contingent on funding and ethics approval, and electronic health record linkage of vital status and episodes of NHS care.

ELIGIBILITY:
Inclusion Criteria:

* History of hospital attendance or hospitalisation for COVID-19, confirmed by a clinical diagnosis, laboratory test e.g. PCR and/or a radiological test e.g. CT chest or chest X-ray
* Age 18 years or more
* Capacity to provide written informed consent
* Able to comply with study procedures

Exclusion Criteria:

* Contra-indication to CMR e.g. severe claustrophobia, metallic foreign body
* Lack of informed consent
* Women who are pregnant, breast-feeding or of child-bearing potential without a negative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers who have attended or admitted to hospital for COVID-19 and meet the eligibility criteria described
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The primary cardiac outcome is the proportion of patients with a diagnosis of myocardial inflammation (myocarditis). | 28 days after discharge from hospital
  Myocardial inflammation (or myocarditis) will be revealed by cardiovascular magnetic resonance imaging (MRI) according to contemporary guidelines including the modified Lake Louise Criteria. The endotypes of myocardial injury are 1) myocardial inflammation due to 1.1) viral myocarditis, 1.2) ischaemia, or 1.3) stress (Takotsubo) cardiomyopathy, 2) myocardial infarction, 3) indeterminate, or 4) none. The final diagnosis will be a consensus-based determination by an expert panel. This information will provide insights into the incidence, nature, time-course and clinical significance of cardiovascular involvement in patients with COVID-19. The clinical significance of our findings will be assessed through associations with patient reported outcome measures (PROMS) and health outcomes in the longer term.
The primary cardio-pulmonary outcome is the proportion of patients with thrombosis | 28 days after discharge from hospital
  Thrombosis of the right heart, pulmonary arteries and left heart will be determined contrast-enhanced CT chest, angiography and MRI.

SECONDARY OUTCOMES:
Myocardial injury | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess mechanisms using circulating biomarkers of cardiac injury, high sensitivity troponin I (ng/L) and its change over time from baseline.
Myocardial stress | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess the significance of myocardial injury by measuring circulating concentrations of NTproBNP (pg/mL) and its change over time from baseline.
Systemic inflammation | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess systemic inflammation by measurement of the peak circulating concentration of C-reactive protein (mg/dL) and its change over time.
Vascular injury | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess vascular injury/inflammation by measurement of the peak circulating concentration of IL-6 (pg/mL) and its change over time.
Endothelial activation and haemostasis | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess endothelial injury by immunoassay measurement of the peak circulating concentration of VWF:ag (IU/dL) and its change over time. Other measures of haemostasis will also be measured.
Fibrin lysis | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess fibrin lysis by measurement of the peak circulating concentration of fibrin D-dimer (IU/dL) and its change over time.
Coagulation | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess coagulation by measurement of Activated Partial Thromboplastin Time (APTT) in seconds. Other measures of coagulation will also be measured.
Platelet count | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess platelet count (n/microlitre), minimum value (thrombocytopaenia) and change over time.
Renal function | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Assess renal function using urine albumin:creatinine ratio and its change over time. Other measures of renal function/injury will also be assessed.
Quantify myocardial perfusion as a measure of coronary microvascular function | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Stress perfusion MRI will provide quantitative assessments of myocardial perfusion (ml/min/g) and classify perfusion abnormalities according to other MRI findings e.g. scar, inflammation and coronary artery disease as revealed by CT coronary angiography.
Association of the primary outcome according to a prior history of cardiovascular disease or no history of prior cardiovascular disease. | 28 days after discharge from hospital, > 1 year post discharge (average 18-22 months)
  Imaging for coronary disease, PTE and lung pathology will be correlated with NHS clinical data on prior history of cardiovascular disease.
Patient reported outcome measures (PROMS) - health status | 1 year
  Health status, well being and function will be prospectively assessed using prespecified PROMS : EuroQOL EQ-5D-5L score. Other measures of health status will also be assessed.
PROMS - functional capacity | 1 year
  Patient reported functional activity using the Duke Activity Status Index (DASI), measured by the score generated from the questionnaire (https://www.mdcalc.com/duke-activity-status-index-dasi)

OTHER OUTCOMES:
Cardiovascular science - vascular biology | 1 year
  Exploratory study to help better understand the cardiovascular pathophysiology of COVID-19. The outcome is endothelial function in of isolated arterioles from gluteal biopsy. Endothelial function will be the (Emax, % vasorelaxation to acetylcholine in a pre-constricted arteriole). Other measures of vascular function will also be assessed.
Cardiovascular science - mathematical modelling | 1 year
  Exploratory study to help better understand the cardiac biomechanical implications of COVID-19. The outcome measure will be myocardial stiffness (Cauchy stress, kPa). The sub-studies will involve using mathematical modelling and, relatedly, statistical emulation. The models will also include the coronary/pulmonary circulation.
Cardiovascular science - pathology | 1 year
  The pathogenesis of SARS-CoV-2 will be examined using histopathology techniques. The outcome is SARS-CoV-2 viral protein or RNA identified in cardiovascular cells.
Health outcomes (serious adverse events) | 20 years
  Health outcomes as measured by the occurrence of serious adverse events (SAE) quantified by 1) rehospitalisation and 2) death. These events will be identified in the longer term using electronic record linkage to health records held by government and the National Health Service.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MBChB/PhD, Principal Investigator — University of Glasgow / NHS Greater Glasgow & Clyde
Locations (3):
- United Kingdom (3):
  - Royal Alexandra Hospital, Paisley, Renfrewshire
  - Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow

REFERENCES:
- [Background] Guzik TJ, Mohiddin SA, Dimarco A, Patel V, Savvatis K, Marelli-Berg FM, Madhur MS, Tomaszewski M, Maffia P, D'Acquisto F, Nicklin SA, Marian AJ, Nosalski R, Murray EC, Guzik B, Berry C, Touyz RM, Kreutz R, Wang DW, Bhella D, Sagliocco O, Crea F, Thomson EC, McInnes IB. COVID-19 and the cardiovascular system: implications for risk assessment, diagnosis, and treatment options. Cardiovasc Res. 2020 Aug 1;116(10):1666-1687. doi: 10.1093/cvr/cvaa106. PMID 32352535
- [Background] Cosyns B, Lochy S, Luchian ML, Gimelli A, Pontone G, Allard SD, de Mey J, Rosseel P, Dweck M, Petersen SE, Edvardsen T. The role of cardiovascular imaging for myocardial injury in hospitalized COVID-19 patients. Eur Heart J Cardiovasc Imaging. 2020 Jul 1;21(7):709-714. doi: 10.1093/ehjci/jeaa136. PMID 32391912
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Derived] Sykes R, Morrow AJ, Mangion K, McConnachie A, McIntosh A, Roditi G, Peng L, Rooney C, Scott K, Stobo DB, Berry C, Church C, Bayes H; CISCO-19 investigators. Radiological abnormalities persist following COVID-19 and correlate with impaired health-related quality of life: a prospective cohort study of hospitalised patients. BMJ Open Respir Res. 2025 Feb 10;12(1):e001985. doi: 10.1136/bmjresp-2023-001985. PMID 39929549
- [Derived] Sykes RA, Neves KB, Alves-Lopes R, Caputo I, Fallon K, Jamieson NB, Kamdar A, Legrini A, Leslie H, McIntosh A, McConnachie A, Morrow A, McFarlane RW, Mangion K, McAbney J, Montezano AC, Touyz RM, Wood C, Berry C. Vascular mechanisms of post-COVID-19 conditions: Rho-kinase is a novel target for therapy. Eur Heart J Cardiovasc Pharmacother. 2023 Jun 2;9(4):371-386. doi: 10.1093/ehjcvp/pvad025. PMID 37019821
- [Derived] Sykes R, Morrow AJ, McConnachie A, Kamdar A, Bagot C, Bayes H, Blyth KG, Briscoe M, Bulluck H, Carrick D, Church C, Corcoran D, Delles C, Findlay I, Gibson VB, Gillespie L, Grieve D, Barrientos PH, Ho A, Lang NN, Lowe DJ, Lennie V, MacFarlane P, Mayne KJ, Mark P, McIntosh A, McGeoch R, McGinley C, Mckee C, Nordin S, Payne A, Rankin A, Robertson KE, Ryan N, Roditi GH, Sattar N, Stobo DB, Allwood-Spiers S, Touyz R, Veldtman G, Weeden S, Watkins S, Welsh P, Wereski R, Mangion K, Berry C. Adjudicated myocarditis and multisystem illness trajectory in healthcare workers post-COVID-19. Open Heart. 2023 Feb;10(1):e002192. doi: 10.1136/openhrt-2022-002192. PMID 36822817
- [Derived] Morrow AJ, Sykes R, McIntosh A, Kamdar A, Bagot C, Bayes HK, Blyth KG, Briscoe M, Bulluck H, Carrick D, Church C, Corcoran D, Findlay I, Gibson VB, Gillespie L, Grieve D, Hall Barrientos P, Ho A, Lang NN, Lennie V, Lowe DJ, Macfarlane PW, Mark PB, Mayne KJ, McConnachie A, McGeoch R, McGinley C, McKee C, Nordin S, Payne A, Rankin AJ, Robertson KE, Roditi G, Ryan N, Sattar N, Allwood-Spiers S, Stobo D, Touyz RM, Veldtman G, Watkins S, Weeden S, Weir RA, Welsh P, Wereski R; CISCO-19 Consortium; Mangion K, Berry C. A multisystem, cardio-renal investigation of post-COVID-19 illness. Nat Med. 2022 Jun;28(6):1303-1313. doi: 10.1038/s41591-022-01837-9. Epub 2022 May 23. PMID 35606551
- [Derived] Mangion K, Morrow A, Bagot C, Bayes H, Blyth KG, Church C, Corcoran D, Delles C, Gillespie L, Grieve D, Ho A, Kean S, Lang NN, Lennie V, Lowe DJ, Kellman P, Macfarlane PW, McConnachie A, Roditi G, Sykes R, Touyz RM, Sattar N, Wereski R, Wright S, Berry C. The Chief Scientist Office Cardiovascular and Pulmonary Imaging in SARS Coronavirus disease-19 (CISCO-19) study. Cardiovasc Res. 2020 Dec 1;116(14):2185-2196. doi: 10.1093/cvr/cvaa209. PMID 32702087
- See also: Glasgow Clinical Trials Unit — https://www.glasgowctu.org/Home
- See also: Chief Scientist Office, Scottish Government - Rapid Research in Covid-19 (RARC-19) — https://www.cso.scot.nhs.uk/covidcalloutcome/